CLINICAL TRIAL: NCT02502097
Title: A Randomized Placebo-Controlled Study to Assess the Efficacy and Safety of AF-219, a P2X3 Receptor Antagonist, in Subjects With Idiopathic Pulmonary Fibrosis (IPF) With Persistent Cough
Brief Title: A Study of Gefapixant (AF-219/MK-7264) in Participants With Idiopathic Pulmonary Fibrosis (IPF) With Persistent Cough (MK-7264-016)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Afferent Pharmaceuticals, Inc., a subsidiary of Merck & Co., Inc. (Rahway, New Jersey USA) (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 7264-016; AF-219-016 (Other: Afferent Pharmaceuticals); MK-7264-016 (Other: Merck Protocol Number)
Record Dates: First submitted 2015-07-16; First posted 2015-07-20 (Estimated); Results first posted 2021-05-26 (Actual); Last update posted 2021-05-26 (Actual); Status verified 2021-04

CONDITIONS: Idiopathic Pulmonary Fibrosis; Cough
MeSH Terms: conditions — Idiopathic Pulmonary Fibrosis; Cough | interventions — Gefapixant

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Gefapixant>Placebo Pre-Amendment 3 (Experimental): Gefapixant 50 mg twice daily (BID) for 10 days, then 150 mg BID for 4 days in Period 1, followed by a 14-21 day washout period, then placebo BID for 14 days in Period 2
  Interventions: Drug: Gefapixant; Other: Placebo
- Placebo>Gefapixant Pre-Amendment 3 (Experimental): Placebo BID for 14 days in Period 1, followed by a 14-21 day washout period, then gefapixant 50 mg BID for 10 days, then 150 mg for 4 days in Period 2
  Interventions: Drug: Gefapixant; Other: Placebo
- Gefapixant>Placebo Post-Amendment 3 (Experimental): Gefapixant 50 mg twice daily (BID) for 14 days in Period 1, followed by a 14-21 day washout period, then placebo BID for 14 days in Period 2
  Interventions: Drug: Gefapixant; Other: Placebo
- Placebo>Gefapixant Post-Amendment 3 (Experimental): Placebo BID for 14 days in Period 1, followed by a 14-21 day washout period, then gefapixant 50 mg BID for 14 days in Period 2
  Interventions: Drug: Gefapixant; Other: Placebo

INTERVENTIONS:
Drug: Gefapixant — Gefapixant 50 mg tablet, administered by mouth
  Other Names: AF-219; MK-7264
Other: Placebo — Matching placebo to gefapixant, tablet administered by mouth

SUMMARY:
A randomized, double-blind, placebo-controlled, crossover, dose escalation study of gefapixant (AF-219) in participants with Idiopathic Pulmonary Fibrosis (IPF) with persistent cough.

DETAILED DESCRIPTION:
Prior to Amendment 3, participants were randomized to receive either placebo twice daily (BID) for 14 days during Period 1 followed by gefapixant 50 mg BID for 10 days then gefapixant 150 mg BID for 4 days BID during Period 2; or gefapixant 50 mg BID for 10 days then gefapixant 150 mg BID for 4 days during Period 1, followed by placebo BID for 14 days during Period 2. Each period was separated by a 14 to 21-day washout period.

During Amendment 3, participants were randomized to receive either placebo BID for 14 days during Period 1 followed by gefapixant 50 mg BID for 14 days during Period 2; or gefapixant 50 mg BID for 14 days during Period 1, followed by placebo BID for 14 days during Period 2. Each period was separated by a 14 to 21-day washout period.

ELIGIBILITY:
Inclusion Criteria:

* Idiopathic pulmonary fibrosis diagnosis based upon the American Thoracic Society (ATS)/ European Respiratory Society (ERS)/Japanese Respiratory Society (JRS)/ Latin American Thoracic Society (ALAT) IPF 2011 guideline
* Life expectancy of greater than 6 months
* Stable medical condition (IPF) for at least 4 weeks
* Self-reported history of troublesome daily cough for more than 8 weeks
* Score of ≥ 40mm on the Cough Severity Visual Analogue Scale (VAS) at Screening
* Women of child-bearing potential must use 2 forms of acceptable birth control method from Screening through the Follow-Up Visit
* Male subjects and their partners of child-bearing potential must use 2 methods of acceptable birth control from Screening until 3 months after the last dose of study drug
* Written informed consent
* Willing and able to comply with all aspects of the protocol

Exclusion Criteria:

* Current smoker (i.e., within the last 30 days).
* Initiation of treatment with an ACE-inhibitor within 4 weeks prior to the Baseline Visit (Day 0) or during the study
* History of upper and/or lower respiratory tract infection within 4 weeks of the Baseline Visit (Day 0)
* History of opioid use for treatment of cough within 1 week of the Baseline Visit (Day 0)
* Requiring prohibited medications
* Body mass index (BMI) <18 kg/m^2 or ≥ 40 kg/m^2
* History or symptoms of renal disease or renal obstructive disease
* History of concurrent malignancy or recurrence of malignancy within 2 years prior to Screening (not including subjects with <3 excised basal cell carcinomas)
* History of a diagnosis of drug or alcohol dependency or abuse within approximately the last 3 years
* Any condition possibly affecting drug absorption (e.g., gastrectomy, gastroplasty, any type of bariatric surgery, vagotomy, or bowel resection)
* Recent history of stroke or transient ischemic attack (within 6 months prior to Screening) not due to trauma, repaired vascular malformation, or aneurysm
* Screening systolic blood pressure (SBP) >160 mm Hg or a diastolic blood pressure (DBP) >90 mm Hg
* QTc interval >450 milliseconds in males, >470 milliseconds in females
* Significantly abnormal laboratory tests at Screening
* Breastfeeding
* Treatment with an investigational drug or biologic within 30 days preceding the first dose of study medication or plans to take another investigational drug or biologic within 30 days of study completion
* Blood donation within 56 days or plasma donation within 7 days prior to dosing
* Other severe, acute, or chronic medical or psychiatric condition or laboratory abnormality that may increase the risk associated with trial participation or investigational product administration or may interfere with the interpretation of trial results

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2015-08-26 (Actual); Primary Completion 2016-07-01 (Actual); Study Completion 2016-07-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC

IPD SHARING:
Plan to Share IPD: Yes
http://engagezone.msd.com/doc/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- [Derived] Martinez FJ, Afzal AS, Smith JA, Ford AP, Li JJ, Li Y, Kitt MM; Chronic Cough in IPF Study Group. Treatment of Persistent Cough in Subjects with Idiopathic Pulmonary Fibrosis (IPF) with Gefapixant, a P2X3 Antagonist, in a Randomized, Placebo-Controlled Clinical Trial. Pulm Ther. 2021 Dec;7(2):471-486. doi: 10.1007/s41030-021-00162-9. Epub 2021 Jun 21. PMID 34152585

RESULTS

PARTICIPANT FLOW:
Period: Period 1
Arm/Group | Gefapixant>Placebo Pre-Amendment 3 | Placebo>Gefapixant Pre-Amendment 3 | Gefapixant>Placebo Post-Amendment 3 | Placebo>Gefapixant Post-Amendment 3
Started | 4 | 3 | 22 | 22
Completed | 4 | 3 | 21 | 22
Not Completed | 0 | 0 | 1 | 0
Not completed — Adverse Event | 0 | 0 | 1 | 0
Period: Wash Out Period
Arm/Group | Gefapixant>Placebo Pre-Amendment 3 | Placebo>Gefapixant Pre-Amendment 3 | Gefapixant>Placebo Post-Amendment 3 | Placebo>Gefapixant Post-Amendment 3
Started | 4 | 3 | 21 | 22
Completed | 4 | 2 | 20 | 21
Not Completed | 0 | 1 | 1 | 1
Not completed — Adverse Event | 0 | 1 | 1 | 1
Period: Period 2
Arm/Group | Gefapixant>Placebo Pre-Amendment 3 | Placebo>Gefapixant Pre-Amendment 3 | Gefapixant>Placebo Post-Amendment 3 | Placebo>Gefapixant Post-Amendment 3
Started | 4 | 2 | 20 | 21
Completed | 4 | 2 | 19 | 21
Not Completed | 0 | 0 | 1 | 0
Not completed — Adverse Event | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Gefapixant>Placebo Pre-Amendment 3 | Placebo>Gefapixant Pre-Amendment 3 | Gefapixant>Placebo Post-Amendment 3 | Placebo>Gefapixant Post-Amendment 3 | Total
Number analyzed (Participants) | 4 | 3 | 22 | 22 | 51
Age, Continuous [Mean (Standard Deviation); unit: Years] | 73.0 (5.35) | 66.7 (0.53) | 69.0 (9.43) | 70.0 (5.06) | 69.6 (7.17)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 1 | 3 | 6 | 11
  Male | 3 | 2 | 19 | 16 | 40
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 1 | 1
  Not Hispanic or Latino | 4 | 3 | 22 | 21 | 50
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0
  White | 4 | 3 | 22 | 21 | 50
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Mixed Model of Repeated Measures (MMRM) Change From Baseline in Awake Objective Cough Frequency (Periods 1 & 2 Combined)
Description: Cough monitoring was conducted for 24 hours while awake, at pre-dose on Day 0 (baseline), and after administration of the study drug on Day 7 and Day 14 in Periods 1 and 2. The cough frequency is the coughs/hour over each 24-hour period. Awake objective cough frequency was analyzed using Mixed Effect Model for Repeated Measures (MMRM) to evaluate the results of the 2-period cross-over study. Baseline cough frequency was derived from the cough monitoring performed at the beginning of each treatment period while the post-treatment cough frequency was derived from the cough monitoring performed at the end of the dosing period. A negative change indicates a decrease in cough frequency, while a positive change indicates an increase in cough frequency.
Time Frame: Baseline (Day 0), Day 7, and Day 14 (Period 1 and Period 2)
Population: The analysis population includes all randomized participants who had a baseline and at least 1 post-baseline frequency values, were enrolled into the study under protocol amendment 3, and had otherwise complied with the protocol without any major protocol deviations. Participants enrolled prior to protocol amendment 3 were not included in the efficacy analysis.
Measure: Least Squares Mean (Standard Error); unit: Coughs/hour
Groups:
- Gefapixant: Gefapixant 50 mg BID for 14 days during 1 of 2 periods
- Placebo: Placebo BID for 14 days during 1 of 2 periods
Arm/Group | Gefapixant | Placebo
Number analyzed (Participants) | 39 | 39
Coughs/hour
  Day 7 | -9.1 (2.7) | -6.6 (2.7)
  Day 14 | -6.6 (4.5) | -5.8 (4.4)
Statistical Analysis 1: Comparison: Gefapixant vs Placebo; Test type: Superiority — MMRM model uses the change from baseline as the dependent variable and includes the period, treatment group (Gefapixant 50 mg, Placebo), visit (Day 7 and Day 14 at each Period), all interactions terms as fixed factors, and baseline as a covariate; p = 0.5096, Mixed Models Analysis; Mean Difference (Final Values) = -2.5, 95% CI 2-sided [-10.1 to 5.1] — LS mean difference Day 7
Statistical Analysis 2: Comparison: Gefapixant vs Placebo; Test type: Superiority — [test comment as in outcome 1, analysis 1]; p = 0.8983, Mixed Models Analysis; Mean Difference (Final Values) = -0.8, 95% CI 2-sided [-13.4 to 11.8] — LS mean difference Day 14

2. Primary Outcome: Awake Objective Cough Frequency (Periods 1 & 2 Combined)
Description: Cough monitoring was conducted for 24 hours while awake, at pre-dose on Day 0 (baseline), and after administration of the study drug on Day 7 and Day 14 in Periods 1 and 2. The cough frequency is the coughs/hour over each 24-hour period. Awake objective cough frequency was defined as the total number of cough events during the monitoring period the participant was awake divided by the total duration for the monitoring period the participant was awake. Baseline cough frequency was derived from the cough monitoring performed at the beginning of each treatment period while the post-treatment cough frequency was derived from the cough monitoring performed at the end of the dosing period.
Time Frame: Baseline (Day 0), Day 7, and Day 14 (Period 1 and Period 2)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Coughs/hour
Arm/Group | Gefapixant | Placebo
Number analyzed (Participants) | 39 | 39
Coughs/hour
  Baseline | 46.2 (43.06) | 48.0 (55.17)
  Day 7: number analyzed (Participants) | 36 | 37
  Day 7 | 37.1 (46.52) | 41.8 (50.11)
  Day 14: number analyzed (Participants) | 36 | 38
  Day 14 | 39.4 (57.67) | 41.9 (44.37)

3. Primary Outcome: Change From Baseline of Awake Objective Cough Frequency (Periods 1 & 2 Combined)
Description: Cough monitoring was conducted for 24 hours while awake, at pre-dose on Day 0 (baseline), and after administration of the study drug on Day 7 and Day 14 in Periods 1 and 2. The cough frequency is the coughs/hour over each 24-hour period. Awake objective cough frequency was defined as the total number of cough events during the monitoring period the participant was awake divided by the total duration for the monitoring period the participant was awake. Baseline cough frequency was derived from the cough monitoring performed at the beginning of each treatment period while the post-treatment cough frequency was derived from the cough monitoring performed at the end of the dosing period. A negative value indicates a decrease in cough frequency.
Time Frame: Baseline (Day 0), Day 7, and Day 14 (Period 1 and Period 2)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Coughs/hour
Arm/Group | Gefapixant | Placebo
Number analyzed (Participants) | 39 | 39
Coughs/hour
  Day 7: number analyzed (Participants) | 36 | 37
  Day 7 | -8.8 (21.81) | -6.6 (13.36)
  Day 14: number analyzed (Participants) | 36 | 38
  Day 14 | -5.9 (36.76) | -5.7 (19.63)

4. Primary Outcome: Percent Change From Baseline of Awake Objective Cough Frequency (Periods 1 & 2 Combined)
Description: Awake objective cough frequency was defined as the total number of cough events during the monitoring period the participant was awake divided by the total duration for the monitoring period the participant was awake. Percent change from baseline in awake objective cough frequency (0-6 hours after the morning dose) was reported at each dosing interval. Percent change in awake cough frequency = 100 X (post treatment cough frequency - baseline cough frequency) divided by the baseline cough frequency. A negative value indicates a decrease in cough frequency.
Time Frame: Baseline (Day 0), Day 7, and Day 14 (Period 1 and Period 2)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Percent change
Arm/Group | Gefapixant | Placebo
Number analyzed (Participants) | 39 | 39
Percent change
  Day 7: number analyzed (Participants) | 36 | 37
  Day 7 | -18.2 (50.06) | -14.1 (31.14)
  Day 14: number analyzed (Participants) | 36 | 38
  Day 14 | -11.9 (60.00) | 6.6 (58.83)

5. Secondary Outcome: MMRM Analysis of Change From Baseline in Awake Objective Cough Frequency (Period 1)
Description: Awake objective cough frequency was defined as the total number of cough events during the monitoring period the participant was awake divided by the total duration for the monitoring period the participant was awake. Change from Baseline in awake cough frequency = post-treatment awake cough frequency - Baseline awake cough frequency. A negative value indicates a decrease in cough frequency. A positive value indicates an increase in cough frequency. Baseline cough frequency was derived from the cough monitoring performed at the beginning of each treatment period while the post-treatment cough frequency was derived from the cough monitoring performed at the end of the dosing period. Awake objective cough frequency for Period 1 was analyzed for using MMRM to evaluate the results of the 2-period cross-over study. The derived change measured at each dose were the repeated measures.
Time Frame: Baseline (Day 0), Day 7, and Day 14 (Period 1)
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Coughs/hour
Arm/Group | Gefapixant | Placebo
Number analyzed (Participants) | 19 | 20
Coughs/hour
  Day 7 | -15.6 (4.0) | -11.9 (3.7)
  Day 14 | -14.9 (6.6) | -13.1 (6.1)
Statistical Analysis 1: Comparison: Gefapixant vs Placebo; Test type: Superiority — [test comment as in outcome 1, analysis 1]; p = 0.5005, Mixed Models Analysis; Mean Difference (Final Values) = -3.7, 95% CI 2-sided [-14.6 to 7.2] — LS means difference Day 7
Statistical Analysis 2: Comparison: Gefapixant vs Placebo; Test type: Superiority — [test comment as in outcome 1, analysis 1]; p = 0.8382, Mixed Models Analysis; Mean Difference (Final Values) = -1.8, 95% CI 2-sided [-19.8 to 16.1] — LS means difference Day 14

6. Secondary Outcome: MMRM Analysis of Change From Baseline in Awake Objective Cough Frequency (Period 2)
Description: Awake objective cough frequency was defined as the total number of cough events during the monitoring period the participant was awake divided by the total duration for the monitoring period the participant was awake. Change from baseline in awake cough frequency = post-treatment awake cough frequency - Baseline awake cough frequency. A negative value indicates a decrease in cough frequency. A positive value indicates an increase in cough frequency. Baseline cough frequency was derived from the cough monitoring performed at the beginning of each treatment period while the post-treatment cough frequency was derived from the cough monitoring performed at the at the end of the dosing period. Awake objective cough frequency for Period 2 was analyzed using MMRM to evaluate the results of the 2-period cross-over study. The derived change measured at each dose were the repeated measures.
Time Frame: Baseline (Day 0), Day 7, and Day 14 (Period 2)
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Coughs/hour
Arm/Group | Gefapixant | Placebo
Number analyzed (Participants) | 20 | 19
Coughs/hour
  Day 7 | -2.7 (3.7) | -1.3 (3.8)
  Day 14 | 1.7 (6.2) | 1.5 (6.4)
Statistical Analysis 1: Comparison: Gefapixant vs Placebo; Test type: Superiority — [test comment as in outcome 1, analysis 1]; p = 0.8008, Mixed Models Analysis; Mean Difference (Final Values) = -1.3, 95% CI 2-sided [-11.9 to 9.2] — LS means difference Day 7
Statistical Analysis 2: Comparison: Gefapixant vs Placebo; Test type: Superiority — [test comment as in outcome 1, analysis 1]; p = 0.9805, Mixed Models Analysis; Mean Difference (Final Values) = 0.2, 95% CI 2-sided [-17.6 to 18.0] — LS means difference Day 14

7. Secondary Outcome: Responder Analysis of Awake Cough Frequency at Day 7 (Periods 1 & 2 Combined)
Description: Awake objective cough frequency was defined as the total number of cough events during the monitoring period the participant was awake divided by the total duration for the monitoring period the participant was awake. The number of participants that met responder criteria for ≥70%, ≥50%, ≥30%, and ≥20% change (reduction) from baseline levels in 24-hour awake cough frequency was reported (Period 1 and Period 2 combined) at Day 7.
Time Frame: Day 7 (Period 1 and Period 2)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Gefapixant | Placebo
Number analyzed (Participants) | 36 | 37
Participants
  Day 7: >= 70% reduction | 1 | 1
  Day 7: >= 50% reduction | 8 | 5
  Day 7: >= 30% reduction | 19 | 11
  Day 7: >= 20% reduction | 22 | 13

8. Secondary Outcome: Responder Analysis of Awake Cough Frequency at Day 14 (Periods 1 & 2 Combined)
Description: Awake objective cough frequency was defined as the total number of cough events during the monitoring period the participant was awake divided by the total duration for the monitoring period the participant was awake. The number of participants that met responder criteria for ≥70%, ≥50%, ≥30%, and ≥20% change (reduction) from baseline levels in 24-hour awake cough frequency was reported (Period 1 and Period 2 combined) at Day 14.
Time Frame: Day 14 (Period 1 and Period 2)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Gefapixant | Placebo
Number analyzed (Participants) | 36 | 38
Participants
  Day 14: >= 70% reduction | 3 | 1
  Day 14: >= 50% reduction | 11 | 3
  Day 14: >= 30% reduction | 18 | 10
  Day 14: >= 20% reduction | 19 | 15

9. Secondary Outcome: MMRM Analysis of Change From Baseline 24-hour Objective Cough Frequency (Periods 1 & 2 Combined)
Description: 24-hour objective cough frequency = total number of coughs during the monitoring period divided by the total duration for the monitoring period. A negative value indicates a decrease in cough frequency. A positive value indicates an increase in cough frequency. 24-hour objective cough frequency was analyzed using MMRM to evaluate the results of the 2-period cross-over study. The derived change measured at each dose were the repeated measures.
Time Frame: Baseline (Day 0), Day 7, and Day 14 (Period 1 and Period 2)
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Coughs/hour
Arm/Group | Gefapixant | Placebo
Number analyzed (Participants) | 39 | 39
Coughs/hour
  Day 7 | -7.1 (1.7) | -4.7 (1.7)
  Day 14 | -2.5 (3.9) | -4.0 (3.8)
Statistical Analysis 1: Comparison: Gefapixant vs Placebo; Test type: Superiority — [test comment as in outcome 1, analysis 1]; p = 0.3279, Mixed Models Analysis; Mean Difference (Final Values) = -2.4, 95% CI 2-sided [-7.1 to 2.4] — LS means difference Day 7
Statistical Analysis 2: Comparison: Gefapixant vs Placebo; Test type: Superiority — [test comment as in outcome 1, analysis 1]; p = 0.7772, Mixed Models Analysis; Mean Difference (Final Values) = 1.5, 95% CI 2-sided [-9.2 to 12.3] — LS means difference Day 14

10. Secondary Outcome: MMRM Analysis of Change From Baseline in 24-hour Objective Cough Frequency (Period 1)
Description: 24-hour objective cough frequency = total number of coughs during the monitoring period divided by the total duration for the monitoring period. A negative value indicates a decrease in cough frequency. A positive value indicates an increase in cough frequency. 24-hour objective cough frequency for Period 1 was analyzed using MMRM to evaluate the results of the 2-period cross-over study. The derived change measured at each dose were the repeated measures.
Time Frame: Baseline (Day 0), Day 7, and Day 14 (Period 1)
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Coughs/hour
Arm/Group | Gefapixant | Placebo
Number analyzed (Participants) | 19 | 20
Coughs/hour
  Day 7 | -11.8 (2.5) | -8.5 (2.3)
  Day 14 | -9.1 (5.6) | -10.1 (5.2)
Statistical Analysis 1: Comparison: Gefapixant vs Placebo; Test type: Superiority — [test comment as in outcome 1, analysis 1]; p = 0.3493, Mixed Models Analysis; Mean Difference (Final Values) = -3.2, 95% CI 2-sided [-10.1 to 3.6] — LS means difference Day 7
Statistical Analysis 2: Comparison: Gefapixant vs Placebo; Test type: Superiority — [test comment as in outcome 1, analysis 1]; p = 0.8952, Mixed Models Analysis; Mean Difference (Final Values) = 1.0, 95% CI 2-sided [-14.3 to 16.3] — LS means difference Day 14

11. Secondary Outcome: MMRM Analysis of Change From Baseline in 24-hour Objective Cough Frequency (Period 2)
Description: 24-hour objective cough frequency = total number of coughs during the monitoring period divided by the total duration for the monitoring period. A negative value indicates a decrease in cough frequency. A positive value indicates an increase in cough frequency. 24-hour objective cough frequency for Period 2 was analyzed using MMRM to evaluate the results of the 2-period cross-over study. The derived change measured at each dose were the repeated measures.
Time Frame: Baseline (Day 0), Day 7, and Day 14 (Period 2)
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Coughs/hour
Arm/Group | Gefapixant | Placebo
Number analyzed (Participants) | 20 | 19
Coughs/hour
  Day 7 | -2.4 (2.3) | -0.9 (2.4)
  Day 14 | 4.1 (5.3) | 2.1 (5.5)
Statistical Analysis 1: Comparison: Gefapixant vs Placebo; Test type: Superiority — [test comment as in outcome 1, analysis 1]; p = 0.6597, Mixed Models Analysis; Mean Difference (Final Values) = -1.5, 95% CI 2-sided [-8.1 to 5.2] — LS means difference Day 7
Statistical Analysis 2: Comparison: Gefapixant vs Placebo; Test type: Superiority — [test comment as in outcome 1, analysis 1]; p = 0.7880, Mixed Models Analysis; Mean Difference (Final Values) = 2.1, 95% CI 2-sided [-13.1 to 17.2] — LS means difference Day 14

12. Secondary Outcome: 24-hour Objective Cough Frequency (Periods 1 & 2 Combined)
Description: 24-hour objective cough frequency = total number of coughs during the monitoring period divided by the total duration for the monitoring period.
Time Frame: Baseline (Day 0), Day 7, and Day 14 (Period 1 and Period 2)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Coughs/hour
Arm/Group | Gefapixant | Placebo
Number analyzed (Participants) | 39 | 39
Coughs/hour
  Baseline | 33.6 (33.39) | 35.5 (39.99)
  Day 7: number analyzed (Participants) | 36 | 37
  Day 7 | 26.4 (33.46) | 30.5 (39.09)
  Day 14: number analyzed (Participants) | 36 | 38
  Day 14 | 30.6 (47.27) | 31.2 (34.19)

13. Secondary Outcome: Change From Baseline of 24-hour Cough Frequency (Periods 1 & 2 Combined)
Description: as for outcome 9
Time Frame: Baseline (Day 0), Day 7, and Day 14 (Period 1 and Period 2)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Coughs/hour
Arm/Group | Gefapixant | Placebo
Number analyzed (Participants) | 40 | 40
Coughs/hour
  Day 7: number analyzed (Participants) | 36 | 37
  Day 7 | -6.8 (13.76) | -4.5 (7.78)
  Day 14: number analyzed (Participants) | 36 | 38
  Day 14 | -2.0 (30.47) | -4.0 (16.79)

14. Secondary Outcome: Percent Change From Baseline of 24-hour Cough Frequency (Periods 1 & 2 Combined)
Description: 24-hour objective cough frequency = total number of coughs during the monitoring period divided by the total duration for the monitoring period. Percent change in cough frequency = 100 X (post treatment cough frequency - baseline cough frequency) divided by the baseline cough frequency. A negative value indicates a decrease in cough frequency. A positive value indicates an increase in cough frequency.
Time Frame: Baseline (Day 0), Day 7, and Day 14 (Period 1 and Period 2)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Percent change
Arm/Group | Gefapixant | Placebo
Number analyzed (Participants) | 40 | 40
Percent change
  Day 7: number analyzed (Participants) | 36 | 37
  Day 7 | -20.4 (49.10) | -14.6 (28.97)
  Day 14: number analyzed (Participants) | 36 | 38
  Day 14 | -9.4 (59.22) | -9.7 (64.24)

15. Secondary Outcome: MMRM Analysis of Change From Baseline in Sleep Cough Frequency (Periods 1 & 2 Combined)
Description: Sleep Objective Cough Frequency = Total number of cough events during the monitoring period the participant is asleep divided by the total duration (in hours) for the monitoring period the participant is asleep. 24-hour sound recordings were collected with a digital recording device. A negative result indicates a decrease in cough frequency, while a positive result indicates an increase in cough frequency. Sleep cough frequency was analyzed using MMRM to evaluate the results of the 2-period cross-over study. The derived change measured at each dose were the repeated measures.
Time Frame: Baseline (Day 0), Day 7, and Day 14 (Period 1 and Period 2)
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Coughs/hour
Arm/Group | Gefapixant | Placebo
Number analyzed (Participants) | 38 | 38
Coughs/hour
  Day 7 | -1.8 (1.3) | 0.8 (1.3)
  Day 14 | 3.3 (3.4) | 0.6 (3.3)
Statistical Analysis 1: Comparison: Gefapixant vs Placebo; Test type: Superiority — [test comment as in outcome 1, analysis 1]; p = 0.1856, Mixed Models Analysis; Mean Difference (Final Values) = -2.5, 95% CI 2-sided [-6.3 to 1.3] — LS mean difference Day 7
Statistical Analysis 2: Comparison: Gefapixant vs Placebo; Test type: Superiority — [test comment as in outcome 1, analysis 1]; p = 0.5658, Mixed Models Analysis; Mean Difference (Final Values) = 2.7, 95% CI 2-sided [-6.6 to 12.1] — LS mean difference Day 14

16. Secondary Outcome: MMRM Analysis of Change From Baseline in Cough Visual Analog Scale (VAS) (Periods 1 & 2 Combined)
Description: Cough VAS is scored from 0 to 100 using a 10 mm visual analogue scale with 0 at 0mm and 100 at 10mm with 0 (no cough) and 100 (most severe cough). Baseline cough VAS is defined as average of screening and baseline cough VAS. A negative result indicates a decrease in cough frequency, while a positive result indicates an increase in cough frequency. Cough VAS was analyzed using MMRM to evaluate the results of the 2-period cross-over study. The derived change measured at each dose were the repeated measures.
Time Frame: Baseline (Day 0), Day 7, and Day 14 (Period 1 and Period 2)
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Score on a scale
Arm/Group | Gefapixant | Placebo
Number analyzed (Participants) | 39 | 40
Score on a scale
  Day 7 | -16.3 (3.3) | -8.2 (3.2)
  Day 14 | -14.3 (4.0) | -8.5 (4.0)
Statistical Analysis 1: Comparison: Gefapixant vs Placebo; Test type: Superiority — [test comment as in outcome 1, analysis 1]; p = 0.0847, Mixed Models Analysis; Mean Difference (Final Values) = -8.0, 95% CI 2-sided [-17.2 to 1.1] — LS mean difference Day 7
Statistical Analysis 2: Comparison: Gefapixant vs Placebo; Test type: Superiority — [test comment as in outcome 1, analysis 1]; p = 0.3083, Mixed Models Analysis; Mean Difference (Final Values) = -5.8, 95% CI 2-sided [-17.0 to 5.4] — LS mean difference Day 14

17. Secondary Outcome: MMRM Analysis of Change From Baseline in Cough Quality of Life Questionnaire (CQLQ) (Periods 1 & 2 Combined)
Description: CQLQ is a 28-item scale that has 4 possible responses: 1 = strongly disagree; 2 = disagree; 3 = agree; 4 = strongly agree. Subjects were instructed to circle only 1 response. The total CQLQ score is the sum of the individual item scores; the lowest possible score is 28 and the highest 112. Low CQLQ scores for both total and the 6 domains indicate less impact of cough on health-related quality of life. A negative result indicates a decrease in cough impact on quality of life. CQLQ was analyzed using MMRM to evaluate the results of the 2-period cross-over study. The derived change measured at each dose were the repeated measures.
Time Frame: Baseline (Day 0), Day 7, and Day 14 (Period 1 and Period 2)
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Score on a scale
Arm/Group | Gefapixant | Placebo
Number analyzed (Participants) | 40 | 40
Score on a scale
  Day 7 | -2.3 (1.2) | -0.3 (1.2)
  Day 14 | 0.2 (1.2) | 0.3 (1.2)
Statistical Analysis 1: Comparison: Gefapixant vs Placebo; Test type: Superiority — [test comment as in outcome 1, analysis 1]; p = 0.2290, Mixed Models Analysis; Mean Difference (Final Values) = -2.0, 95% CI 2-sided [-5.3 to 1.3] — LS mean difference Day 7
Statistical Analysis 2: Comparison: Gefapixant vs Placebo; Test type: Superiority — [test comment as in outcome 1, analysis 1]; p = 0.9794, Mixed Models Analysis; Mean Difference (Final Values) = -0.0, 95% CI 2-sided [-3.5 to 3.4] — LS mean difference Day 14

18. Secondary Outcome: MMRM Analysis of Change From Baseline in Total Daily Cough Severity Diary (CSD) Score (Periods 1 & 2 Combined)
Description: The daily CSD Score is calculated using the daily CSD instrument, a 7-item, disease specific, patient-reported outcome measure with a recall period of "today" (the current day). The measure evaluates frequency of cough (3 items); intensity of cough (2 items); and sleep disruption due to cough (2 items). Each of these 7 items is rated on an 11-point scale, ranging from 0 (best) to 10 (worst), with higher scores indicating greater severity. The total daily CSD score is the sum of these 7 item scores (Min=0, Max=70). Baseline CSD score = average of CSD scores at screening and baseline. A negative result indicates a decrease in cough severity, while a positive result indicates an increase in cough severity. CSD was analyzed using MMRM to evaluate the results of the 2-period cross-over study. The derived change measured at each dose were the repeated measures.
Time Frame: Baseline (Day 0), Week 1, and Week 2 (Period 1 and Period 2)
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Score on a scale
Arm/Group | Gefapixant | Placebo
Number analyzed (Participants) | 40 | 40
Score on a scale
  Week 1: number analyzed (Participants) | 36 | 32
  Week 1 | -1.4 (0.2) | -0.4 (0.2)
  Week 2: number analyzed (Participants) | 36 | 31
  Week 2 | -1.7 (0.2) | -0.7 (0.3)
Statistical Analysis 1: Comparison: Gefapixant vs Placebo; Test type: Superiority — [test comment as in outcome 1, analysis 1]; p = 0.0009, Mixed Models Analysis; Mean Difference (Final Values) = -1.0, 95% CI 2-sided [-1.5 to -0.4] — LS mean difference Week 1
Statistical Analysis 2: Comparison: Gefapixant vs Placebo; Test type: Superiority — [test comment as in outcome 1, analysis 1]; p = 0.0050, Mixed Models Analysis; Mean Difference (Final Values) = -1.0, 95% CI 2-sided [-1.7 to -0.3] — LS mean difference Week 2

19. Secondary Outcome: MMRM Analysis of Change From Baseline in University of California San Diego Shortness of Breath Questionnaire (UCSD SOBQ) (Periods 1 & 2 Combined)
Description: UCSD SOBQ is a 24-point item scale to assess shortness of breath questionnaire that has a 6-point scale ranging from 0 to 5 (0 = "not at all", to 5 = "maximal or unable to do because of breathlessness". Lowest possible score is 0 and the highest possible score is 120. The higher the score the more out of breath the participant is reporting. A negative value indicates less breathlessness. UCSD SOBQ was analyzed using MMRM to evaluate the results of the 2-period cross-over study. The derived change measured at each dose were the repeated measures.
Time Frame: Baseline (Day 0), Day 7, and Day 14 (Period 1 and Period 2)
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Score on a scale
Arm/Group | Gefapixant | Placebo
Number analyzed (Participants) | 40 | 40
Score on a scale
  Day 7 | -3.9 (1.9) | -1.0 (1.9)
  Day 14: number analyzed (Participants) | 39 | 39
  Day 14 | -2.4 (1.9) | 1.6 (1.9)
Statistical Analysis 1: Comparison: Gefapixant vs Placebo; Test type: Superiority — [test comment as in outcome 1, analysis 1]; p = 0.2938, Mixed Models Analysis; Mean Difference (Final Values) = -2.8, 95% CI 2-sided [-8.2 to 2.5] — LS mean difference Day 7
Statistical Analysis 2: Comparison: Gefapixant vs Placebo; Test type: Superiority — [test comment as in outcome 1, analysis 1]; p = 0.1319, Mixed Models Analysis; Mean Difference (Final Values) = -4.0, 95% CI 2-sided [-9.2 to 1.2] — LS mean difference Day 14

20. Secondary Outcome: MMRM Analysis of Change From Baseline in Cough Borg CR10 Scale Score (Periods 1 & 2 Combined)
Description: The Borg 10 scale assesses post-treatment breathlessness during perceived exertion while exercising. The scale ranges from 0 to 10 where 0 = nothing at all, 1 = very weak, 3 = moderate, 5 = strong, 7 = very strong, 10 = extremely strong. The lowest possible score is 0 and the highest possible score is 10. A negative value indicates less breathlessness. Cough Borg CR10 was analyzed using MMRM to evaluate the results of the 2-period cross-over study. The derived change measured at each dose were the repeated measures.
Time Frame: Baseline (Day 0), Day 7, and Day 14 (Period 1 and Period 2)
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Score on a scale
Arm/Group | Gefapixant | Placebo
Number analyzed (Participants) | 40 | 40
Score on a scale
  Day 7 | -0.5 (0.3) | 0.1 (0.3)
  Day 14: number analyzed (Participants) | 39 | 39
  Day 14 | -0.1 (0.4) | 0.3 (0.4)
Statistical Analysis 1: Comparison: Gefapixant vs Placebo; Test type: Superiority; p = 0.2175, Mixed Models Analysis; Mean Difference (Final Values) = -0.6, 95% CI 2-sided [-1.5 to 0.4] — LS mean difference Day 7
Statistical Analysis 2: Comparison: Gefapixant vs Placebo; Test type: Superiority; p = 0.5312, Mixed Models Analysis; Mean Difference (Final Values) = -0.3, 95% CI 2-sided [-1.4 to 0.7] — LS mean difference Day 14

21. Secondary Outcome: Percentage of Participants With Borg CR10 Perception of Breathless Value ≥5 (Periods 1 & 2 Combined)
Description: The Borg 10 scale assesses post-treatment breathlessness during perceived exertion while exercising. The scale ranges from 0 to 10 where 0 = nothing at all, 1 = very weak, 3 = moderate, 5 = strong, 7 = very strong, 10 = extremely strong. The lowest possible score is 0 and the highest possible score is 10. The percentage of participants with Borg CR10 perception of breathless value ≥5 was assessed.
Time Frame: Baseline (Day 0), Day 7, and Day 14 (Period 1 and Period 2)
Population: The analysis population includes all randomized participants who received at least 1 dose of study drug. Two participants that had missing values for Day 14 were excluded.
Measure: Number; unit: Percent of Participants
Arm/Group | Gefapixant | Placebo
Number analyzed (Participants) | 48 | 48
Percent of Participants
  Day 7 | 41.67 | 43.75
  Day 14 | 50.00 | 43.75

22. Secondary Outcome: Patient's Global Impression of Change (PGIC) Day 7 (Periods 1 & 2 Combined)
Description: PGIC is the participant self-reported overall improvement of cough following administration of study drug. The PGIC has a 7-point rating scale of "very much improved", "much improved", 'minimally improved", "no change", "minimally worse", "much worse" and "very much worse".
Time Frame: Day 7 (Period 1 and Period 2)
Population: as for outcome 1
Measure: Number; unit: Participants
Arm/Group | Gefapixant | Placebo
Number analyzed (Participants) | 40 | 40
Participants
  Very much improved | 3 | 1
  Much improved | 14 | 5
  Minimally improved | 12 | 10
  No change | 7 | 18
  Minimally worse | 2 | 4
  Much worse | 0 | 1
  Very much worse | 1 | 1

23. Secondary Outcome: Patient's Global Impression of Change (PGIC) Day 15 (Periods 1 & 2 Combined)
Description: as for outcome 22
Time Frame: Day 15 (Period 1 and Period 2)
Population: as for outcome 1
Measure: Number; unit: Participants
Arm/Group | Gefapixant | Placebo
Number analyzed (Participants) | 40 | 38
Participants
  Very much improved | 5 | 4
  Much improved | 16 | 8
  Minimally improved | 8 | 5
  No change | 5 | 16
  Minimally worse | 4 | 3
  Much worse | 1 | 2
  Very much worse | 0 | 0

24. Secondary Outcome: Clinician's Global Impression of Change (CGIC) Day 15 (Periods 1 & 2 Combined)
Description: CGIC is the clinician's-reported overall improvement of participant's cough following administration of study drug. The CGIC has a 7-point rating scale of "very much improved", "much improved", 'minimally improved", "no change", "minimally worse", "much worse" and "very much worse".
Time Frame: Day 15 (Period 1 and Period 2)
Population: as for outcome 1
Measure: Number; unit: Participants
Arm/Group | Gefapixant | Placebo
Number analyzed (Participants) | 40 | 38
Participants
  Very much improved | 7 | 3
  Much improved | 11 | 4
  Minimally improved | 13 | 6
  No change | 4 | 18
  Minimally worse | 2 | 5
  Much worse | 2 | 1
  Very much worse | 0 | 0

25. Secondary Outcome: Taste Acceptability Questionnaire: Number of Participants That Were Likely to Take Study Medication For At Least Six Months
Description: At the end of the treatment period, participants were asked "How likely would you be to take this medication for at least 6 months?" The degree of taste acceptability was measured on a scale of "extremely unlikely", "unlikely", "neither", "likely" and "extremely likely."
Time Frame: After last treatment, up to Day 15 (Period 1 and Period 2)
Population: as for outcome 1
Measure: Number; unit: Participants
Arm/Group | Gefapixant | Placebo
Number analyzed (Participants) | 40 | 38
Participants
  Extremely unlikely | 2 | 1
  Unlikely | 4 | 2
  Neither | 5 | 4
  Likely | 8 | 12
  Extremely likely | 21 | 19

26. Secondary Outcome: Taste Acceptability Questionnaire: Number of Participants That Were Likely to Take Study Medication For At Least One Year
Description: At the end of the treatment period, the participant was asked "How likely would you be to take this medication for at least one year?" The degree of taste acceptability was measured on a scale of "extremely unlikely", "unlikely", "neither", "likely" and "extremely likely."
Time Frame: After last treatment, up to Day 15 (Period 1 and Period 2)
Population: as for outcome 1
Measure: Number; unit: Participants
Arm/Group | Gefapixant | Placebo
Number analyzed (Participants) | 40 | 38
Participants
  Extremely unlikely | 3 | 1
  Unlikely | 3 | 2
  Neither | 5 | 4
  Likely | 11 | 13
  Extremely likely | 18 | 18

27. Other Pre Specified Outcome: Pre-dose Baseline of Awake Objective Cough Frequency
Description: Awake objective cough frequency was defined as the total number of cough events during the monitoring period the participant was awake divided by the total duration for the monitoring period the participant was awake. Baseline cough frequency was derived from the cough monitoring performed at the beginning of each treatment period.
Time Frame: Baseline (Day 0) (Period 1 and Period 2)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Coughs/hour
Arm/Group | Gefapixant | Placebo
Number analyzed (Participants) | 40 | 38
Coughs/hour
  Period 1: number analyzed (Participants) | 19 | 20
  Period 1 | 50.2 (29.50) | 56.1 (71.68)
  Period 2: number analyzed (Participants) | 20 | 19
  Period 2 | 42.5 (53.42) | 39.4 (29.19)

28. Other Pre Specified Outcome: Pre-dose Baseline 24-hour Objective Cough Frequency (Periods 1 & 2 Combined)
Description: 24-hour objective cough frequency = total number of coughs during the monitoring period divided by the total duration for the monitoring period. Baseline 24-hour cough frequency in Periods 1 and 2 was evaluated based on the participant's randomized group (gefapixant or placebo).
Time Frame: Baseline (Day 0) (Period 1 and Period 2)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Coughs/hour
Arm/Group | Gefapixant | Placebo
Number analyzed (Participants) | 39 | 39
Coughs/hour | 33.6 (33.39) | 35.5 (39.99)

29. Other Pre Specified Outcome: Pre-dose Baseline of 24-hour Objective Cough Frequency (Period 1)
Description: 24-hour objective cough frequency = total number of coughs during the monitoring period divided by the total duration for the monitoring period. Baseline 24-hour cough frequency for Period 1 was evaluated based on the participant's randomized group (gefapixant or placebo).
Time Frame: Baseline (Day 0) (Period 1)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Coughs/hour
Arm/Group | Gefapixant | Placebo
Number analyzed (Participants) | 19 | 20
Coughs/hour | 36.1 (22.18) | 42.5 (51.52)

30. Other Pre Specified Outcome: Pre-dose Baseline of 24-hour Objective Cough Frequency (Period 2)
Description: 24-hour objective cough frequency = total number of coughs during the monitoring period divided by the total duration for the monitoring period. Baseline 24-hour objective cough frequency for Period 2 was evaluated based on the participant's randomized group (gefapixant or placebo).
Time Frame: Baseline (Day 0) (Period 2)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Coughs/hour
Arm/Group | Gefapixant | Placebo
Number analyzed (Participants) | 20 | 19
Coughs/hour | 31.1 (41.84) | 28.1 (21.52)

31. Other Pre Specified Outcome: Pre-dose Baseline Sleep Cough Frequency
Description: Sleep Objective Cough Frequency = Total number of cough events during the monitoring period the participant is asleep divided by the total duration (in hours) for the monitoring period the participant is asleep. 24-hour sound recordings were collected with a digital recording device. Baseline sleep cough frequency was evaluated based on the participant's randomized group (gefapixant or placebo).
Time Frame: Baseline (Day 0)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Coughs/hour
Arm/Group | Gefapixant | Placebo
Number analyzed (Participants) | 38 | 38
Coughs/hour | 8.1 (20.83) | 8.5 (21.26)

32. Other Pre Specified Outcome: Pre-dose Baseline Cough VAS (Periods 1 & 2 Combined)
Description: Cough VAS is scored from 0 to 100 using a 10 mm visual analogue scale with 0 at 0mm and 100 at 10mm with 0 (no cough) and 100 (most severe cough). Baseline cough VAS was defined as average of screening and baseline cough VAS.
Time Frame: Baseline (Day 0) (Period 1 and Period 2)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Gefapixant | Placebo
Number analyzed (Participants) | 39 | 40
Score on a scale | 56.0 (24.03) | 53.9 (22.80)

33. Other Pre Specified Outcome: Pre-dose Baseline Cough CQLQ (Periods 1 & 2 Combined)
Description: CQLQ is a 28-item scale that has 4 possible responses: 1 = strongly disagree; 2 = disagree; 3 = agree; 4 = strongly agree. Subjects were instructed to circle only 1 response. The total CQLQ score is the sum of the individual item scores; the lowest possible score is 28 and the highest 112. Low CQLQ scores for both total and the 6 domains indicate less impact of cough on health-related quality of life. Baseline cough CQLQ was evaluated based on the participant's randomized group (gefapixant or placebo).
Time Frame: Baseline (Day 0) (Period 1 and Period 2)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Gefapixant | Placebo
Number analyzed (Participants) | 40 | 40
Score on a scale | 56.5 (13.26) | 56.8 (11.25)

34. Other Pre Specified Outcome: Pre-dose Baseline Cough Severity CSD (Periods 1 & 2 Combined)
Description: The daily CSD Score is calculated using the daily CSD instrument, a 7-item, disease specific, patient-reported outcome measure with a recall period of "today" (the current day). The measure evaluates frequency of cough (3 items); intensity of cough (2 items); and sleep disruption due to cough (2 items). Each of these 7 items is rated on an 11-point scale, ranging from 0 (best) to 10 (worst), with higher scores indicating greater severity. The total daily CSD score is the sum of these 7 item scores (Min=0, Max=70). Baseline CSD score = average of CSD scores at screening and baseline.
Time Frame: Baseline (Day 0) (Period 1 and Period 2)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Gefapixant | Placebo
Number analyzed (Participants) | 36 | 32
Score on a scale | 4.5 (1.75) | 4.1 (2.04)

35. Other Pre Specified Outcome: Pre-dose Baseline of UCSD SOBQ (Periods 1 & 2 Combined)
Description: UCSD SOBQ is a 24-point item scale to assess shortness of breath questionnaire that has a 6-point scale ranging from 0 to 5 (0 = "not at all", to 5 = "maximal or unable to do because of breathlessness". Lowest possible score is 0 and the highest possible score is 120. The higher the score the more out of breath the participant is reporting. Baseline of UCSD SOBQ was evaluated based on the participant's randomized group (gefapixant or placebo).
Time Frame: Baseline (Day 0) (Period 1 and Period 2)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Gefapixant | Placebo
Number analyzed (Participants) | 40 | 40
Score on a scale | 58.0 (26.06) | 57.1 (24.63)

36. Other Pre Specified Outcome: Pre-dose Baseline of Cough Borg CR10 Scale Score (Periods 1 & 2 Combined)
Description: The Borg 10 scale assesses post-treatment breathlessness during perceived exertion while exercising. The scale ranges from 0 to 10 where 0 = nothing at all, 1 = very weak, 3 = moderate, 5 = strong, 7 = very strong, 10 = extremely strong. The lowest possible score is 0 and the highest possible score is 10. The baseline of cough Borg CR10 was evaluated based on the participant's randomized group (gefapixant or placebo).
Time Frame: Baseline (Day 0) (Period 1 and Period 2)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Gefapixant | Placebo
Number analyzed (Participants) | 40 | 40
Score on a scale | 4.4 (3.08) | 3.9 (2.56)

ADVERSE EVENTS:
Time Frame: Up to 63 days (9 weeks)
Description: Analysis population includes all participants who received at least one dose of study drug.
Groups:
- Placebo: Participants received placebo BID for 14 days
- Gefapixant 50 mg: Participants received gefapixant 50 mg BID for 10 or 14 days
- Gefapixant 150 mg: Participants received gefapixant 150 mg BID for 4 days
Arm/Group | Placebo | Gefapixant 50 mg | Gefapixant 150 mg
Serious Adverse Events (participants affected / at risk) | 3/45 | 3/47 | 1/4
Other Adverse Events (participants affected / at risk) | 12/45 | 39/47 | 3/4
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=45) | Gefapixant 50 mg (N=47) | Gefapixant 150 mg (N=4)
Atrial fibrillations (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Palpitations (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Chest pain (General disorders) | 0 (0) | 1 (1) | 0 (0)
Bronchitis (Infections and infestations) | 1 (1) | 1 (1) | 1 (1)
Pneumonia (Infections and infestations) | 2 (2) | 0 (0) | 0 (0)
Dysponea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Interstitial Lung Disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=45) | Gefapixant 50 mg (N=47) | Gefapixant 150 mg (N=4)
Diarrhoea (Gastrointestinal disorders) | 2 (2) | 3 (3) | 0 (0)
Hypoaesthesia oral (Gastrointestinal disorders) | 0 (0) | 4 (5) | 0 (0)
Paraesthesia oral (Gastrointestinal disorders) | 0 (0) | 4 (6) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 5 (5) | 0 (0)
Respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (1) | 3 (3) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Ageusia (Nervous system disorders) | 0 (0) | 11 (14) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 4 (4) | 0 (0)
Dysgeusia (Nervous system disorders) | 1 (1) | 25 (28) | 0 (0)
Hypogeusia (Nervous system disorders) | 0 (0) | 5 (6) | 0 (0)
Pollakiuria (Renal and urinary disorders) | 1 (1) | 4 (4) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 6 (7) | 6 (7) | 0 (0)
Rales (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
No data collected as part of this study will be utilized in any written work, including publications, without the written consent of Sponsor.